CLINICAL TRIAL: NCT01613274
Title: The Effect of Gum Chewing on Bowel Motility in Post-operative Colon Resection Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCBM
Record Dates: First submitted 2012-06-03; First posted 2012-06-07 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Colon Resection
Keywords: colon resection
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gum chewing (Experimental): Chewing mint flavored sugarless gum for 10-20 minutes three times a day following colon resection.
  Interventions: Other: gum chewing
- no gum chewing (Placebo Comparator): no gum chewing
  Interventions: Other: no gum chewing

INTERVENTIONS:
Other: gum chewing — gum chewing three times a day for up to 20 minutes
  Arms: Gum chewing
Other: no gum chewing — no gum chewing
  Arms: no gum chewing

SUMMARY:
The purpose of this study is to determine if chewing mint-flavored sugarless gum after colon resection surgery decrease the time to first flatus, bowel movement and length of stay in the hospital.

DETAILED DESCRIPTION:
Post-operative colon resection patients experience decreased bowel motility, which may cause pain, nausea/ vomiting, impaired nutritional intake, and abdominal distention. Return of bowel function is a strong determinant in length of hospital stay. There are small studies that have shown that chewing gum post-operatively may enhance bowel motility thus minimizing complications and decreasing length of hospital stay. The purpose of this research study is to determine the effect of gum chewing on bowel motility as measured by time to first flatus, bowel movement and length of stay in patients following a colon resection.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to Unit 2600
2. Age 18-100 years of age
3. Alert and oriented
4. Post-operative open or laparoscopic colon resection
5. English speaking.

Exclusion Criteria:

1. Confused, or with cognitive disabilities that render the patient unable to answer questions about bowel motility.
2. Admitted to any other unit except 2600
3. Use of an epidural catheter for pain control post-operatively
4. Documented history of irritable bowel syndrome
5. Colostomy (new or old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Time to first flatus | Every 4 hours following surgery until discharge, which is an average of 5 days

SECONDARY OUTCOMES:
Time to first bowel movement | Every 4 hours following surgery until discharge, which is an average of 5 days
Length of stay in days | Patients will be followed until discharge, which is an average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Sabo, RN Mn CNS-BC, Principal Investigator — United Hospital
Locations (1):
- United Hospital, Saint Paul, Minnesota, United States